CLINICAL TRIAL: NCT02396316
Title: A Randomized, Double-masked, and Controlled Phase 3 Study to Evaluate the Efficacy, Safety, and Tolerability of Intravitreal Administration of Aflibercept in Japanese Patients With Neovascular Glaucoma
Brief Title: Japanese Phase 3 Study of Aflibercept in Neovascular Glaucoma Patients
Acronym: VEGA
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bayer (Industry)
Collaborators: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 17584
Record Dates: First submitted 2015-03-18; First posted 2015-03-24 (Estimated); Results first posted 2017-07-21 (Actual); Last update posted 2017-09-15 (Actual); Status verified 2017-08

CONDITIONS: Glaucoma, Neovascular
MeSH Terms: conditions — Glaucoma, Neovascular | interventions — aflibercept; salicylhydroxamic acid

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Aflibercept (Experimental): Aflibercept 2 mg Intravitreal (IVT) injection group
  Interventions: Drug: Aflibercept (Eylea, BAY 86-5321)
- Sham Injection (Sham Comparator): Sham injection group
  Interventions: Drug: Sham Injection

INTERVENTIONS:
Drug: Aflibercept (Eylea, BAY 86-5321) — After the first aflibercept IVT injection on Day 1, subjects may receive sham injection at Week 1, and aflibercept injection at Week 5 and/or Week 9 if the re-treatment criteria are met.
  Arms: Aflibercept
Drug: Sham Injection — After the first sham injection on Day 1, subjects may receive aflibercept IVT injection at Week 1, Week 5 and/or Week 9 if re-treatment criteria are met.
  Arms: Sham Injection

SUMMARY:
To assess the efficacy and safety of the administration of aflibercept by intravitreal injection in comparison to sham to control intraocular pressure in patients with neovascular glaucoma.

ELIGIBILITY:
Inclusion Criteria:

* Japanese men and women aged 20 years or older,
* Patients diagnosed as having Neovascular glaucoma (NVG) with neovascularization in the anterior segment (both iris and anterior chamber angle),
* Patients with Intraocular pressure (IOP) higher than 25 mmHg in the study eye due to anterior segment (both iris and anterior chamber angle) neovascularization.

Exclusion Criteria:

* Patients with angle-closure due to conditions other than Neovascular glaucoma
* Patients with a known or suspected ocular or peri-ocular infection,
* Patients with severe intraocular inflammation in the study eye,
* Women who are pregnant, suspected of being pregnant or lactating,
* Patients with known allergy to aflibercept.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2015-04-02 (Actual); Primary Completion 2016-06-16 (Actual); Study Completion 2016-09-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (19):
- Japan (19):
  - Yoshida, Fukui
  - Gifu, Gifu
  - Amagasaki, Hyōgo
  - Himeji, Hyōgo
  - Kobe, Hyōgo
  - Kanazawa, Ishikawa-ken
  - Kawasaki, Kanagawa
  - Sendai, Miyagi
  - Yufu, Oita Prefecture
  - Hirakata, Osaka
  - Suita, Osaka
  - Takatsuki, Osaka
  - Izumo, Shimane
  - Bunkyo-ku, Tokyo
  - Mitaka, Tokyo
  - Ube, Yamaguchi
  - Chūō, Yamanashi
  - Kyoto
  - Osaka

REFERENCES:
- [Derived] Rittiphairoj T, Roberti G, Michelessi M. Anti-vascular endothelial growth factor for neovascular glaucoma. Cochrane Database Syst Rev. 2023 Apr 3;4(4):CD007920. doi: 10.1002/14651858.CD007920.pub4. PMID 37010901
- [Derived] Inatani M, Higashide T, Matsushita K, Miki A, Ueki M, Iwamoto Y, Kobayashi M, Leal S; VEGA Investigators. Intravitreal Aflibercept in Japanese Patients with Neovascular Glaucoma: The VEGA Randomized Clinical Trial. Adv Ther. 2021 Feb;38(2):1116-1129. doi: 10.1007/s12325-020-01579-5. Epub 2020 Dec 16. PMID 33330958

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study was conducted at nineteen study centers in Japan, between 02 April 2015 (first subject first visit) and 06 Sep 2016 (last subject last visit).
Pre-assignment Details: A total of 63 subjects were screened and 54 subjects were randomized into the aflibercept group (N=27) and the sham group (N =27).
Groups:
- Aflibercept 2 mg Intravitreal (IVT) Injection Group: Subjects received intravitreal (IVT) injection of 2 mg (0.05 milliliter [ml] * 40 milligram per milliliter [mg/ml]) aflibercept on Day 1. Then, subjects may receive sham injection at Week 1, and aflibercept injection at Week 5 and/or Week 9 if the re-treatment criteria are met. Re-treatment criteria (subjects could receive aflibercept IVT injection when all the following retreatment criteria were met) :
  * IOP higher than 21mmHg;
  * Incomplete regression of iris neovascularization and;
  * Aflibercept IVT deemed necessary by the investigator.
- Sham Injection Group: Subjects received a sham injection on Day 1. Then, subjects may receive aflibercept injection at Week 1, Week 5 and/or Week 9 if the re-treatment criteria specified in the protocol are met. Re-treatment criteria (subjects could receive aflibercept IVT injection when all the following retreatment criteria were met) :
  * IOP higher than 21mmHg;
  * Incomplete regression of iris neovascularization and;
  * Aflibercept IVT deemed necessary by the investigator.
Period: Overall Study
Arm/Group | Aflibercept 2 mg Intravitreal (IVT) Injection Group | Sham Injection Group
Started | 27 | 27
Treated | 27 | 27
Received Sham Injection at Week 1 | 10 | 0
Received AFL Injection at Week 1 | 0 | 22
Received Active Injection at Week 5 | 4 | 4
Received Active Injection at Week 9 | 2 | 1
Completed | 20 | 22
Not Completed | 7 | 5
Not completed — Physician Decision | 1 | 0
Not completed — Progressive disease | 6 | 3
Not completed — Protocol Violation | 0 | 1
Not completed — Treatment unblinded | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Aflibercept 2 mg Intravitreal (IVT) Injection Group | Sham Injection Group | Total
Number analyzed (Participants) | 27 | 27 | 54
Age, Continuous [Mean (Standard Deviation); unit: Years] | 68.1 (12.7) | 66.2 (13.7) | 67.1 (13.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 4 | 9
  Male | 22 | 23 | 45

OUTCOME MEASURES:

1. Primary Outcome: Change in Intraocular Pressure (IOP) From Baseline to Pre-dose at Week 1
Description: It compared the change in IOP from baseline to pre-dose at Week 1 between the aflibercept group vs the sham group.
Time Frame: From baseline to pre-dose at Week 1
Population: FAS: The Full Analysis Set (FAS) included all randomized subjects who have received any study drug (including sham injection) and had had a baseline and at least one post-baseline IOP measurement on a posterior date. The FAS was analyzed as randomized.
Measure: Mean (Standard Deviation); unit: mmHg
Groups:
- Aflibercept 2 mg Intravitreal (IVT) Injection Group: Subjects received intravitreal (IVT) injection of 2 mg (0.05 ml * 40 mg/ml) aflibercept on Day 1. Then, subjects may receive sham injection at Week 1, and aflibercept injection at Week 5 and/or Week 9 if the re-treatment criteria are met.
  Re-treatment criteria (subjects could receive aflibercept IVT injection when all the following retreatment criteria were met) :
  * IOP higher than 21mmHg;
  * Incomplete regression of iris neovascularization and;
  * Aflibercept IVT deemed necessary by the investigator.
Arm/Group | Aflibercept 2 mg Intravitreal (IVT) Injection Group | Sham Injection Group
Number analyzed (Participants) | 27 | 27
mmHg | -8.5 (8.7) | -4.9 (10.8)
Statistical Analysis 1: Comparison: Aflibercept 2 mg Intravitreal (IVT) Injection Group vs Sham Injection Group; Point estimate, 95% CI and P-value were based on treatment difference of the LS mean changes using an ANCOVA model with treatment group and stage of NVG for randomization as fixed effects, baseline value as covariate. The superiority of aflibercept injection to sham injection was to be established if the upper limit of the two-sided 95% confidence interval for the difference (the aflibercept group minus the sham group) is less than 0; Test type: Superiority or Other; p = 0.0644, ANCOVA; Difference of LS mean change = -4.9, 95% CI 2-sided [-10.2 to 0.3]

2. Secondary Outcome: Percentage of Subjects Who Had Improved Neovascularization of the Iris (NVI) Grade From Baseline to Pre-dose at Week 1
Description: NVI were assessed in the study eye using the NVI grading systems (grade 0 to grade 4). A subject who shows the improvement by at least one grade is considered to be improved. Percentage of subjects who had improved NVI grade was reported.
Time Frame: From baseline to pre-dose at Week 1
Population: FAS
Measure: Number; unit: Percentage of participants
Arm/Group | Aflibercept 2 mg Intravitreal (IVT) Injection Group | Sham Injection Group
Number analyzed (Participants) | 27 | 27
Percentage of participants | 70.4 | 11.5
Statistical Analysis 1: Comparison: Aflibercept 2 mg Intravitreal (IVT) Injection Group vs Sham Injection Group; The point estimate of the treatment difference (the aflibercept group minus the sham group) at Week 1 and its two-sided 95% confidence interval stratified by stage of NVG (as randomized) using Mantel-Haenszel weights; Test type: Superiority or Other; Mantel Haenszel; MH adjusted difference = 59.1, 95% CI 2-sided [37.0 to 81.2]

ADVERSE EVENTS:
Time Frame: Adverse event data were collected after the first dose of study drug and no later than 30 days after the last dose of study drug. AEs from the first dose of study drug until pre-dose at Week 1 were also reported.
Groups:
- Aflibercept 2 mg Intravitreal (IVT) Injection Group: Subjects received intravitreal (IVT) injection of 2 mg (0.05 ml * 40 mg/ml) aflibercept on Day 1. Then, subjects may receive sham injection at Week 1, and aflibercept injection at Week 5 and/or Week 9 if the re-treatment criteria are met.
  Re-treatment criteria (subjects could receive aflibercept IVT injection when all the following retreatment criteria were met) :
  * IOP higher than 21mmHg;
  * Incomplete regression of iris neovascularization and;
  * Aflibercept IVT deemed necessary by the investigator. (AE time frame: from first dose of study drug until 30 days after the last dose of study drug)
- Sham Injection Group: Subjects received a sham injection on Day 1. Then, subjects may receive aflibercept injection at Week 1, Week 5 and/or Week 9 if the re-treatment criteria specified in the protocol are met.
  Re-treatment criteria (subjects could receive aflibercept IVT injection when all the following retreatment criteria were met) :
  * IOP higher than 21mmHg;
  * Incomplete regression of iris neovascularization and;
  * Aflibercept IVT deemed necessary by the investigator. (AE time frame: from first dose of study drug until 30 days after the last dose of study drug)
- Aflibercept 2 mg IVT Injection Group (Till Pre-dose at Week 1): Subjects received IVT injection of 2 mg (0.05 ml * 40 mg/ml) aflibercept on Day 1. Then, subjects may receive sham injection at Week 1, and aflibercept injection at Week 5 and/or Week 9 if the re-treatment criteria are met.
  Re-treatment criteria (subjects could receive aflibercept IVT injection when all the following retreatment criteria were met) :
  * IOP higher than 21mmHg;
  * Incomplete regression of iris neovascularization and;
  * Aflibercept IVT deemed necessary by the investigator. (AE time frame: from the first dose of study drug until pre-dose at Week 1)
- Sham Injection Group (Till Pre-dose at Week 1): Subjects received a sham injection on Day 1. Then, subjects may receive aflibercept injection at Week 1, Week 5 and/or Week 9 if the re-treatment criteria specified in the protocol are met.
  Re-treatment criteria (subjects could receive aflibercept IVT injection when all the following retreatment criteria were met) :
  * IOP higher than 21mmHg;
  * Incomplete regression of iris neovascularization and;
  * Aflibercept IVT deemed necessary by the investigator. (AE time frame: from the first dose of study drug until pre-dose at Week 1)
Arm/Group | Aflibercept 2 mg Intravitreal (IVT) Injection Group | Sham Injection Group | Aflibercept 2 mg IVT Injection Group (Till Pre-dose at Week 1) | Sham Injection Group (Till Pre-dose at Week 1)
Serious Adverse Events (participants affected / at risk) | 3/27 | 3/27 | 0/27 | 0/27
Other Adverse Events (participants affected / at risk) | 10/27 | 12/27 | 6/27 | 7/27
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Aflibercept 2 mg Intravitreal (IVT) Injection Group (N=27) | Sham Injection Group (N=27) | Aflibercept 2 mg IVT Injection Group (Till Pre-dose at Week 1) (N=27) | Sham Injection Group (Till Pre-dose at Week 1) (N=27)
Myocardial ischaemia (Cardiac disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Diabetic retinopathy (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Retinal artery occlusion (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Retinal vein occlusion (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Eating disorder (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Aflibercept 2 mg Intravitreal (IVT) Injection Group (N=27) | Sham Injection Group (N=27) | Aflibercept 2 mg IVT Injection Group (Till Pre-dose at Week 1) (N=27) | Sham Injection Group (Till Pre-dose at Week 1) (N=27)
Conjunctival haemorrhage (Eye disorders) | 2 (2) | 1 (1) | 2 (2) | 0 (0)
Eye pain (Eye disorders) | 0 (0) | 4 (5) | 0 (0) | 1 (1)
Hyphaema (Eye disorders) | 0 (0) | 2 (2) | 0 (0) | 2 (2)
Punctate keratitis (Eye disorders) | 2 (4) | 3 (4) | 2 (2) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Injection site pain (General disorders) | 2 (3) | 1 (1) | 2 (3) | 1 (1)
Procedural pain (Injury, poisoning and procedural complications) | 3 (4) | 0 (0) | 0 (0) | 0 (0)
Intraocular pressure increased (Investigations) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 2 (2) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No